CLINICAL TRIAL: NCT05424211
Title: The Effect Of A Mobile Application-Based Music Intervention On Pain Levels And Analgesic Consumption Following Surgery: A Randomized Controlled Trial
Brief Title: The Effect of Music Therapy on Pain Level and Analgesic Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Acelya Turkmen, PhD, Cukurova University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CU-SBF-AT-03
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-02

CONDITIONS: Orthopedic Surgery; Pain, Postoperative; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Music group (Experimental): the group using the music therapy mobile application
  Interventions: Device: Music Therapy Mobile Application
- control group (No Intervention): the group that received routine care and treatment

INTERVENTIONS:
Device: Music Therapy Mobile Application — The authorities determined by taking consultancy from TÜMATA (Turkish Music Research and Promotion Group) will be uploaded to the mobile application developed by the software specialist. The maqams (Rast, Nihavent and Neva) to be used in the application will be played to the patients 3 times in half an hour at different times of the day via the mobile application. Rast tonality will be played in the morning, nihavent tune will be played at noon and neva tune will be played in the afternoon.
  Arms: Music group

SUMMARY:
Pain is a common condition experienced by patients in long-term health care, rehabilitation and acute situations, due to various surgical interventions and invasive procedures, and postoperative pain is an important symptom experienced by patients during the surgical recovery process. The International Association for the Study of Pain (IASP) defines pain as an unpleasant emotional experience associated with actual or potential tissue damage (Lok, Ibrahim and Sidani 2020; Çavdar and Akyüz 2017; Martin-Saavedra, Vergara-Mendez, Talero-Gutiérrez 2018). Orthopedic surgical interventions are considered to be one of the most painful surgical procedures, and pain control requires a multifaceted approach that includes non-pharmacological techniques (Allred et al. 2010). Music therapy, which is one of the non-traditional treatment methods, is used to reduce pain (Nilson 2008). Music can easily be included in nursing care because it is applied without the physician's request and causes very little legal and ethical concerns (Simcock et al. 2008). However, due to the lack of awareness about the effectiveness of music therapy, it is not often used as an intervention. Inadequate pain control causes a decrease in patient satisfaction and deterioration of the healing process (Lukas 2004). Therefore, this study was planned as a randomized controlled experimental study to determine the effect of music therapy on the pain level of patients undergoing orthopedic surgery.

DETAILED DESCRIPTION:
This study was planned as a randomized controlled experimental study to determine the effect of music therapy on the level of pain after orthopedic surgery. The population of the research will consist of patients who have undergone orthopedic surgery in the orthopedic service of a university hospital. In a similar study in the literature (Tolunay et al. 2018), the number of samples was calculated on the basis of 95% confidence interval, 80% power level, 0.05 error level, 0.84 effect level, considering the pain averages of the experimental and control groups. As a result of the power analysis, at least 19 patients were included in the experimental and control groups, and it was determined that a total of at least 38 patients could form the sample group; however, it was decided to complete the study with a total of 80 patients by assigning 40 patients to each group so that parametric tests could be performed during the data analysis.

Inclusion criteria for the study: Accepting to participate in the study, being over 18 years old, having undergone orthopedic surgery, not having mental and auditory problems, not having chronic pain, being literate.

Exclusion criteria for the study: being younger than 18 years of age, undergoing non-elective orthopedic surgery, coming from the intensive care unit, having mental and auditory problems, chronic pain, illiteracy.

Data will be collected by Patient Information Form, Numerical Scale (NRS) and Short Form.

Implementation of Research:

First stage: All patients who meet the sampling criteria will be informed about the type, purpose and application process of the pre-intervention study, and written and verbal consent will be obtained for participation. In order to prevent individuals from being informed about the interventions, the participants will be randomized to the experimental and control groups according to the period of admission to the hospital. According to the results of randomization, patients will be assigned to the group (experimental group) and the control group. Researchers will maintain the confidentiality of patients' identity and study-related information using serial numbers.

Second stage: After the explanations about the study are made and the necessary written and verbal consent is obtained, a structured information form containing information about socio-demographic variables such as age, gender, education, alcohol and smoking use, chronic disease of all participants will be filled.

Third stage:

Music Therapy Mobile Application: The authorities determined by consulting TÜMATA (Turkish Music Research and Promotion Group) will be uploaded to the mobile application developed by the software specialist. The maqams (Rast, Nihavent and Neva) to be used in the application will be played to the patients 3 times in half an hour at different times of the day via the mobile application. Rast tonality will be played in the morning, nihavent tune will be played at noon and neva tune will be played in the afternoon. Each patient will be given a personal headphone probe to listen to music.

Pain assessment will be done with NRS before and immediately after the application. Routine treatment and care of the patients in the control group will continue.

ELIGIBILITY:
Inclusion Criteria:

Accepting to participate in the study, being over the age of 18, having undergone orthopedic surgery, not having mental and auditory problems, not having chronic pain, being able to read and write

Exclusion Criteria:

Being younger than 18 years of age, undergoing non-elective orthopedic surgery, coming from the intensive care unit, having mental and auditory problems, chronic pain, illiteracy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-05-02 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
The Numerical Rating Scale (NRS) | 1 year
  It starts with the absence of pain (0) on numerical scales and reaches the level of unbearable pain (10-100). Numerical scales are used by patients to facilitate the definition of pain intensity, to facilitate scoring and recording, and to evaluate ceiling and floor effects.

SECONDARY OUTCOMES:
Analgesic consumption amount | 1 year
  The amount of analgesic used by the patients after the surgery will be recorded in the table.

CONTACTS AND LOCATIONS:
Overall Officials: Açelya Türkmen, PhD, Study Chair — Cukurova University
Locations (1):
- Cukurova University, Adana, Sarıcam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No